CLINICAL TRIAL: NCT04514770
Title: Early Versus Late Amniotomy on Labour Induction in Nulliparous Women
Brief Title: Impact of Early Versus Late Amniotomy on Labour Induction in Nulliparous Women After Vaginal Misoprostol
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Elsibai Anter, Lecturer of obstetrics and gynecology, Menoufia Obstetrics and Gynecology Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/2019 OBSGN 27
Record Dates: First submitted 2020-07-28; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Labour Induction
MeSH Terms: interventions — Misoprostol; Amniotomy

STUDY DESIGN:
Intervention Model Description: Group A: Early amniotomy was performed for the participant of the first group at 3 cm cervical dilatation with Kocher's forceps provided the head is well fitted to the cervix. Group B: late amniotomy was performed for the participant of the second group at 7 cm cervical dilatation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early amniotomy (Active Comparator): Group A:
  1. Pregnant women had taken misoprostol (vagiprost vaginal tablet; Adwia Pharmaceutical Company) vaginally as 25 micro gram of misoprostol. It was repeated every 6 hours until three or more uterine contractions of 40 second duration occur over 10 minutes, or when reaching four doses maximum (i.e. 100 micro gram) is reached.
  2. Early amniotomy was performed for the participant of the first group at 3 cementer cervical dilatation with Kocher's forceps provided the head is well fitted to the cervix.
  Interventions: Drug: Misoprostol
- Late amniotomy (Active Comparator): Group B:
  1. Pregnant women had taken misoprostol (vagiprost vaginal tablet; Adwia Pharmaceutical Company) vaginally as 25 micro gram of misoprostol. It was repeated every 6 hours until three or more uterine contractions of 40 second duration occur over 10 minutes, or when reaching four doses maximum (i.e. 100 micro gram) is reached.
  2. late amniotomy was performed for the participant of the second group at 7 cementer cervical dilatation.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — rupture of membrane early and late
  Other Names: Amniotomy

SUMMARY:
Investigation the effect of timing of amniotomy (early versus delayed) after vaginal misoprostol in induced labor.

Condition: induction of labour intervention: eary versus late amniotomy on labour induction after vaginal misoprostol Phase: Not applicable

DETAILED DESCRIPTION:
study type: randomized clinical trial actual enrollment: 140 allocation: Random intervention model: two groups assignment masking: open lebal primary purpose: induction of labour actual study start: May 3, 2019 Primary Completion: January 10, 2020 actual study completion date: March 20, 2020

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women at 36 weeks gestation or more
2. Nullipara
3. singleton fetus
4. cephalic presentation with common medical causes for labour induction e.g. intrauterine fetal growth restriction, post term pregnancy and preeclampsia.

Exclusion Criteria:

1. Macrocosmic babies with estimated fetal weight of more than 4000 gram
2. Previous uterine scars
3. Pre labor premature rupture of fetal membranes
4. Polyhydramnios.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Nulliparous Women
Enrollment: 140 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
successful induction | immediately after intervention
  definition of successful induction is occurrence of vaginal delivery within 24 hours from the beginning of induction
induction-delivery interval | immediately after intervention
  duration of labor and amniotomy delivery interval

SECONDARY OUTCOMES:
misoprostol doses administered | during the intervention
  number of misoprostol doses administered
the need for augmentation of labor | during the intervention
  the need for augmentation of labor by oxytocin and perinatal outcomes included cord prolapse and abnormal FHR changes during labor
intrapartum meconium | during the intervention
  intrapartum meconium passage
Apgar score | during the intervention
  Apgar score less than 7 at 1 and 5 minutes
newborn admission in the neonatal intensive care unit | immediately after intervention
  newborn admission in the neonatal intensive care unit (NICU).

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University hospital, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No